CLINICAL TRIAL: NCT05831397
Title: Extracellular Vesicles as a Diagnostic and Prognostic Biomarker of Neoadjuvant Chemotherapy (NAC) in Breast Cancer Patients.
Brief Title: Extracellular Vesicles in Breast Cancer Patientsin Undergone Neoadjuvant Chemotherapy
Status: Recruiting | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Principal Investigator, Fabio Corsi, Professor, Istituti Clinici Scientifici Maugeri SpA
Other Study IDs: 2540
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Breast cancer patients candidate for neoadjuvant chemotherapy: Female patients diagnosed with breast cancer, at any TNM stage, who are candidate to neoadjuvant treatment.
- Healty control: Control group (sex and age matched): healthy volunteers, not affected by breast cancer (with negative mammography, breast ultrasound or breast examination within 12 months of the study enrolment).

SUMMARY:
Extracellular vesicles (EVs) are lipid bilayer-delimited particles, naturally released from the cells and mediators of intercellular cross-talk. In breast cancer (BC), EVs seem to be involved in the tumor microenvironment's shaping, in cancer cells invasion and in the set-up of metastasis.

Clinical studies have provided initial evidence that EVs may have a prognostic and predictive value in breast cancer. Considering their presence in body fluids and their minimally invasive assessment through blood sampling, EVs could be liquid biopsy-derived biomarkers. Their quantification could be a complex challenge, requiring complicated and time-consuming pre-analytical procedures of EVs isolation.

A new method for the detection of tumor-derived-EVs associated proteins is based on the use of Single Molecule Array (SiMoA), a digital ELISA technology able to detect and quantify extremely low concentrations of target proteins or particles.

The aim of this study is to evaluate how this new technology can allow the quantification EVs plasma levels in patients affected by BC, providing useful diagnostic and prognostic information about the efficacy of the neoadjuvant treatment.

DETAILED DESCRIPTION:
This is a prospective, observational, monocentric and no profit study. The study involves the analysis of plasma from patients with breast cancer to quantify and characterize tumor-derived EVs at specific disease stages, and to evaluate the efficacy of the neoadjuvant treatment.

BC patients will be consequently included, at any TNM stage, undergoing neoadjuvant chemotherapy referring to an EUSOMA-accredited Breast Unit.

Patients will be divided into two groups, as follows:

* Population 1: female patients diagnosed with breast cancer, at any TNM stage, who are candidate to neoadjuvant treatment.
* Population 2: a control group of sex and age matched healthy volunteers, not affected by breast cancer (with negative mammography, breast ultrasound or breast examination within 12 months of the study enrolment).

For each BC patient, 4 blood samples will be collected at established time-points and plasma will be isolated. Blood samples will be collected as follows: the first sample (T0) before the first chemotherapy infusion; the second sample (T1) before the second chemotherapy infusion (Day 21); the third sample (T2) after the last chemotherapy infusion and before the surgical treatment (between 21 and 42 days after the last chemotherapy infusion); fourth and last sample 1 month after surgery (T3).

A new SiMoA assay, based on the use of anti-CD63 and anti-CD9 antibodies, will be used to quantify EVs directly from plasma without requiring any prior sample processing.

The study will be conducted following the International Conference on Harmonization [ICH] Good Clinical Practice [GCP] guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Signing of a specific informed consent for participation to the study
* Female sex

BC patients:

* Diagnosis of breast cancer
* Any TNM stage
* Indication to neoadjuvant chemotherapy after multidisciplinary discussion

Healthy controls:

• Patients with a negative mammography, breast ultrasound or clinical breast evaluation within 12 months of the study enrolment

Exclusion Criteria:

BC patients:

• Indication to upfront surgery

Healthy controls:

• Diagnosis of breast cancer

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer is gender based
Study Population: * Population 1: female patients diagnosed with breast cancer, at any TNM stage, who are candidate to neoadjuvant treatment.
  * Population 2: a control group of sex and age matched healthy volunteers, not affected by breast cancer (with negative mammography, breast ultrasound or clinical breast examination within 12 months of the study enrolment).
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2021-05-11 (Actual); Primary Completion 2027-12-21 (Estimated); Study Completion 2027-12-21 (Estimated)

PRIMARY OUTCOMES:
EVs levels | 78 months
  Measurement of plasma EVs levels (by Simoa-Elisa) in BC patients at the moment of diagnosis and comparison between EVs concentration in BC patients' and healthy controls.
EVs levels in time | 78 months
  Evaluation of tumor-related EVs as predictive markers of neoadjuvant treatment efficacy in BC patients. This will be conducted comparing EVs level during different collected times

CONTACTS AND LOCATIONS:
Locations (1):
- Istituti Clinici Scientifici Maugeri SpA, Pavia, Lombardy, Italy